CLINICAL TRIAL: NCT04946773
Title: Deep Liver Phenotyping and Immunology Study
Acronym: DELPHI
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 264839; C2195/A27431 (Other Grant/Funding Number: Cancer Research UK); CA30358/A29725 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2021-06-09; First posted 2021-07-01 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma
Keywords: Early Detection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Tissue, blood, urine & bile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignancy Cohort: Patients with hepatic or hepatobiliary malignancy at enrolment
- Control Cohort: Patients with chronic liver disease but no hepatic or hepatobiliary malignancy at enrolment

SUMMARY:
Hepatocellular carcinoma (HCC) and cholangiocarcinoma are the two most common causes of primary liver cancer and HCC is the second highest cause of cancer death worldwide. It is known that most of these cancers occur in patients who already have a liver condition. Despite close monitoring of many patients who have liver disease with regular ultrasound scans, HCC and cholangiocarcinoma are often discovered at a late stage. This is because they rarely cause symptoms until they have reached an advanced stage. Early identification of these cancers would enable more patients to have curative treatments such as surgery or liver transplantation.

The investigators want to collect blood and urine samples as well as small samples of cells directly from the liver. In some cases this will be done using a technique called liver fine needle aspiration. This technique is low risk and has been successfully used in other studies. The investigators will compare samples from patients with cancer to those of patients with other diseases of the liver who are at risk of developing cancer in the future.

The investigators aim to detect changes in the liver, blood, urine and/or bile of patients who have liver conditions that could tell us their risk of a future cancer. These changes could be in the types of white blood cells found within the liver, or, they may be in products secreted by liver cells. In the latter case the liver cells may release small pieces of their DNA that could be detected in the blood. When liver cells are dysfunctional, they may also change the types of metabolic products that they produce, and the investigators may be able to detect these changes in the urine or bile.

DETAILED DESCRIPTION:
The purpose of this study is to perform a characterisation of the cancer predisposing 'field effect' that is associated with hepatic & hepato-biliary malignancy, and, to identify minimally invasive biomarkers that may detect this field effect. This will be achieved through collection of patient samples (Tissue/Blood/Urine/Bile). Comparisons will then be made between patients with hepatic & hepatobiliary cancer and patients with chronic liver disease and also longitudinally in individual patients who either develop or are cured of hepatic & hepato-biliary malignancy during the study. The investigators hope to exploit this knowledge to develop novel biomarker candidates that may ultimately form inputs to a multi-parametric early cancer detection model. The study aims are:

1. Develop a cohort of patients with HCC, cholangiocarcinoma or liver metastases and a cohort of chronic liver disease patients representing all the commonly encountered aetiologies (viral, metabolic, autoimmune and alcohol related liver disease).
2. Collect samples from directly within the non-cancerous liver (FNA liver/biopsy/ablation/resection specimens), blood and urine in addition tumour tissue (resection/biopsy/ablation), bile and bile duct brushings.
3. Flow cytometric & molecular biologic analysis of tissue and peripheral blood and bile.
4. Transcriptomic analysis of cell populations in liver and blood.
5. Genetic & molecular biologic analysis of hepatic and immune cells and secreted products.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years to 75 years.

Malignancy Cohort: extra inclusion criteria - Diagnosed with a malignancy or with clinical suspicion of a malignancy affecting the Liver or Biliary Tree.

Control cohort: extra inclusion criteria

- Patients with confirmed chronic non-malignant hepatobiliary disease.

Additional Inclusion Criteria for Patients Undergoing optional Liver FNA

* Willing to undergo ultrasound guided liver FNA (unless specific contra-indications to the procedure apply).
* Has undergone appropriate clinical imaging of the upper abdomen (US/CT/MRI) within the last 12 months.
* Full blood count (FBC) and coagulation profile (Coag) checked within 30 days prior to FNA procedure (Baseline Visit).

Exclusion Criteria:

* Unable to consent.
* Pregnancy.
* Any concern by the investigator regarding the safe participation of the patient in the study; or investigator's consideration, for any other reason, that a patient is inappropriate for participation in the study.

Additional Exclusion Criteria for Patients Undergoing optional Liver FNA (These criteria will exclude a patient from having FNA as part of the study)

* Significant comorbid medical condition(s) which may in the opinion of the investigator increase the risk of an FNA Liver.
* Coagulopathy - International Normalized Ratio (INR) >1.3, Prothrombin Time (PT) >16 seconds, Platelet count <100 x 10^3/L.
* Known bleeding disorder (e.g. Haemophilia).
* Current use of an oral/injectable anticoagulant medication.
* Current use of an oral antiplatelet agent.
* The presence of ascites.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatology patients treated at a single hospital trust.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2040-10-31 (Estimated); Study Completion 2040-10-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of intra-hepatic and peripheral blood immune cell numbers in Malignancy Cohort and Control Cohort patients. | At study enrolment
  Proportion of immune cell populations relative to total immune cell count measured by single cell RNA sequencing.

SECONDARY OUTCOMES:
Measurement of liver cancer occurrence and all-cause mortality. | 15 years
  Measurement of absolute numbers of liver cancers and deaths in study patients

OTHER OUTCOMES:
Measure safety of fine needle aspiration in cirrhosis | 5 years
  Measurement of absolute numbers of adverse events related to liver fine needle aspiration in study patients with cirrhosis.
Measure tolerability of liver fine needle aspiration | 5 years
  Measure post procedure analgesia dose and duration in patients undergoing liver fine needle aspiration as a study procedure

CONTACTS AND LOCATIONS:
Overall Officials: Rory J Peters, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom